CLINICAL TRIAL: NCT07357961
Title: The Effectiveness of a Theory-driven Behavioral Change Intervention on Sedentary Behavior in Individuals With Coronary Heart Disease: A Randomised Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Elaine Yi Ning Miu, PhD Candidate, Registered Nurse, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CREC_2025.458
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: sedentary behaviour; movement behaviours
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: The intervention is guided by the Temporal Self-Regulation Theory.
Who Masked: Outcomes Assessor
Masking Description: The study employs single masking, where only the outcome assessor is blinded. Due to the nature of the interventions, masking the participants and intervention providers is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to the usual care, which is the same as the control group, participants allocated to the intervention group will receive a 12-week theory-driven behavioural change intervention. The intervention is structured into eight individual sessions, including four face-to-face sessions (45 minutes each) and four telephone sessions (20 minutes each).
  Interventions: Behavioral: A theory-driven behavioural change intervention
- Attention controlled Group (Active Comparator): Participants in the control group will continue to have the usual care and education sessions, consisting of information about healthy lifestyles, except physical activity and sedentary behaviour.
  Interventions: Behavioral: Attentive control group

INTERVENTIONS:
Behavioral: A theory-driven behavioural change intervention — A theory-driven behavioural change intervention is validated by an expert panel including professionals from various fields, such as nurse consultants, a specialty nurse in cardiology, an experienced registered nurse from a cardiac rehabilitation center in a regional hospital, a physiotherapist, and academia, focusing on strengthening intention to change (connected beliefs and temporal valuations), behavioral prepotency, and enhancing the self-regulatory capacity, as guided by the Temporal Self-Regulation Theory, and supplemented with a intervention booklet. The intervention is developed and facilitated by a registered nurse (principal investigator).
  Arms: Intervention group
Behavioral: Attentive control group — Participants in the attention control group will participate in education sessions consisting of information about healthy lifestyles, except physical activity and sedentary behaviour. Activities match the time and attention dedicated by the intervention group. Activities are designed to have no impact on sedentary behaviour and physical activity.
  Arms: Attention controlled Group

SUMMARY:
The objective of this randomised controlled trial is to examine the effectiveness of a theory-driven behavioural change intervention on total sedentary time (primary outcomes), moderate-to-vigorous physical activity time, intention of behavioural change, future time perception, behavioural prepotency, self-regulation capacity, and exercise capacity in individuals with coronary heart disease.

Hypotheses:

Compared to the participants in the control group, participants in the intervention group will demonstrate:

1. Significantly less total sedentary time
2. Significantly improved MVPA time,
3. Significantly better intention of behavioural change,
4. Significantly higher level of behavioural prepotency,
5. Significantly enhanced self-regulation capacity, and
6. Significantly greater future time perception
7. Significantly better exercise capacity at the immediate post-intervention (T1), the 1-month post-intervention (T2), and the 6-month post-intervention (T3).

Participants will:

Participants in the intervention group will participate in a theory-driven behavioural change intervention over three months, comprising four individual face-to-face sessions (45 minutes each) and four individual telephone sessions (20 minutes each), along with the usual care.

Participants in the attention control group will continue to have the usual care, which includes regular follow-up at the cardiac clinic. Education sessions, consisting of information about healthy lifestyles, except physical activity and sedentary behaviour, with the same schedule as the intervention group, will be provided to account for potential attention effects from contacts.

DETAILED DESCRIPTION:
Coronary heart disease is a worldwide health problem and a major contributor to disability, with a high prevalence of 315 million cases globally in 2022. Promoting movement behaviours, which are characterised by having an adequate amount of physical activity and replacing sedentary behaviour with physical activity of all intensities, is beneficial for cardiometabolic health and thus secondary prevention. However, reviews of interventional studies indicate that currently available non-pharmacological interventions are effective in increasing the amount of physical activity, yet limited attention is given to the reduction of sedentary behaviour in current cardiac rehabilitation. Therefore, it is imperative to develop an non-pharmacological intervention targeting sedentary behaviour for adults with coronary heart disease based on the synthesised scientific evidence. The design of the theory-driven behavioural change intervention is based on the findings of our published systematic review and the implications of the qualitative study.

This randomised controlled trial evaluate a theory-driven behavioural change intervention for individuals with coronary heart disease. The objective of the study aims to examine the effectiveness of the intervention in reducing total sedentary time (primary outcome) and improving MVPA, behavioural intentions, future time perception, behavioural prepotency, self-regulation capacity, and exercise capacity in a larger sample.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18 years old and above
2. Diagnosed with coronary heart disease within one year
3. Engaged in MVPA less than 150 minutes per week and a minimum of 8 hours total sedentary time per day, both assessed using the Global Physical Activity Questionnaire
4. Able to communicate in Cantonese
5. Obtained medical clearance for physical activity (no medical contraindications to exercise, including walking)
6. Being able to understand and give informed consent
7. Having telephone access, text messaging services or WhatsApp

Exclusion Criteria:

1. Cannot perform brisk walking exercise
2. Unable to perform PA independently
3. Cognitive impairments, as indicated by an abbreviated mental test score of less than 7
4. Currently enrolled in another clinical trial focusing on limiting SB with/without enhancing PA
5. Doctor-diagnosed psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Total sedentary time | Pre-intervention, post-intervention (within 1 week immediately after intervention), and at 1-month and 6-month follow-ups.
  Total sedentary time (per day) will be measured using the ActiGraph accelerometer (ActiGraph,Pensacola, FL), wGT3X-BT (during participants' waking time over 7 consecutive days, including both weekdays and weekends).

SECONDARY OUTCOMES:
Moderate-to-vigorous physical activity time | Pre-intervention, post-intervention (within 1 week immediately after intervention), and at 1-month and 6-month follow-ups.
  Moderate-to-vigorous physical activity time (per week) will be measured using the ActiGraph accelerometer (ActiGraph, Pensacola, FL), wGT3X-BT (during participants' waking time over seven consecutive days, including both weekdays and weekends).
Self-regulation capacity | Pre-intervention, post-intervention (within 1 week immediately after intervention), and at 1-month and 6-month follow-ups.
  Self-regulation capacity will be measured using the Chinese version of the Brief Self-Control Scale (BSCS).
Behavioural prepotency | Pre-intervention, post-intervention (within 1 week immediately after intervention), and at 1-month and 6-month follow-ups.
  Behavioural prepotency (on both MVPA and SB) will be measured using the Chinese version of the Self-Reported Behavioural Automaticity Index (SRBAI).
Future time perception | Pre-intervention, post-intervention (within 1 week immediately after intervention), and at 1-month and 6-month follow-ups.
  Future time perception will be measured using the Chinese version of the Consideration of Future Consequences Scale (CFCS-14).
Intention of behavioural change | Pre-intervention, post-intervention (within 1 week immediately after intervention), and at 1-month and 6-month follow-ups.
  Intention of behavioural change will be measured using three questions, including (1) I intend to ...; (2) I plan to ...; and (3) It is likely that I will ... Specifically, questions such as "I intend to do at least 150 minutes of MVPA in the coming week" and "I intend to engage in less than 8 hours of total sedentary time per day in the coming week" will be asked, and participants will respond on a 7-point Likert scale ranging from "strongly disagree" to "strongly agree." The sum average will be calculated. Higher scores represent higher intention.
Exercise capacity | Pre-intervention, post-intervention (within 1 week immediately after intervention), and at 1-month and 6-month follow-ups.
  Exercise capacity will be measured using Six-Minute Walk Test, a exercise test that refletsfunctional capacity in daily activity. The test was conducted in a flat, straight, indoor corridor of 30 meters. Participants were instructed to walk back and forth along the corridor, covering as much distance as possible within six minutes, at a self-selected pace, with the option to slow down or rest if necessary. Standardized encouragement was provided at regular intervals. The total distance walked (Six-Minute Walk Distance), measured in meters, was recorded. Heart rate, oxygen saturation, blood pressure, and perceived exertion were monitored before and immediately after the test to ensure participant safety.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Yi Ning Miu, MSc, Principal Investigator — Chinese University of Hong Kong; Ho Yu Cheng, PhD, Study Director — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
The research team does not have plans to proactively or automatically make the individual participant data (IPD) from this study available to other researchers. However, the IPD may be shared upon request, provided that the requesting party has a valid scientific or medical rationale and obtains the necessary approval from the research team.
  Any requests for access to the study's IPD will be reviewed on a case-by-case basis by the research team. Factors that will be considered in evaluating such requests include:
  Scientific merit and validity of the proposed use of the data Qualifications and track record of the requesting researcher or research team Alignment with the original study objectives and participants' consent